CLINICAL TRIAL: NCT05744154
Title: A Multifaceted Intervention to Reduce Low-value Care for Trauma Admissions: Evaluation of Effectiveness in a Pragmatic Cluster Randomized Controlled Trial
Brief Title: Reducing Low-value Care for Trauma Admissions
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Institut national en santé et services sociaux (Unknown); Trauma Association of Canada (Unknown); Health Standards Organisation (Unknown); Choosing Wisely Canada (Unknown); Audit & Feedback Metalab (Unknown); Institut national de la pertinence des actes médicaux (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 113664
Record Dates: First submitted 2023-02-06; First posted 2023-02-24 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Trauma Injury
Keywords: Low-value care; Multifaceted intervention; De-implementation; Trauma system
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Intervention Model Description: We will conduct a parallel arm, pragmatic cluster randomized trial (CRT) embedded in the provincial trauma quality assurance program. As the trial will be based on routinely collected data that are available at no extra cost, we will use a baseline observation period pre-randomization to increase study power. We will randomize at the hospital level because quality programs operate at the local trauma committee level in each hospital. A stepped wedge design will not be used as the minimum one-year roll-out period is unacceptably long for stakeholders and parallel arm CRTs have fewer risks of bias than stepped wedge CRTs. The trial is pragmatic as the intervention will be embedded in the 2023 evaluation cycle of the provincial quality assurance program.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Local trauma committees will not be told explicitly what aspect of the intervention is randomised; they will only be aware that there are two variations of the intervention. Data extractors and analysts will be blinded to group allocation. Due to the nature of the intervention, it will not be possible to blind the investigators to allocation groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Audit & feedback with educational outreach and facilitation (Experimental): The intervention includes: 1) refinement with end users, 2) an A&F report sent to local governing authorities presenting for each practice: performance compared to peers (simple A&F), a summary message indicating if action is required and a list of potential actions, 3) educational materials (a clinical vignette; consequences of the practice; links to practice guidelines, clinical decision rules and shared decision-making tools; a case review tool), 4) virtual educational meetings with the local trauma Medical Director, trauma program manager and data analyst, and 5) two virtual facilitation visits 2 and 4 months after the transmission of the report to support committees in preparing their action plan.
  Interventions: Behavioral: Audit & feedback with educational outreach and facilitation
- Simple audit & feedback (Other): The control arm will receive the quality improvement intervention currently in place in the Québec Trauma Care Continuum (i.e. simple A&F report presenting their performance compared to peers on quality indicators measuring adherence to high-value care and risk-adjusted outcomes) with the addition of quality indicators on low-value care (already planned by provincial authorities for the 2023 evaluation cycle). Simple A&F was chosen for the control because it is standard practice in Québec and in most integrated trauma systems and the effectiveness of A&F for de-implementation has been documented.
  Interventions: Behavioral: Simple audit & feedback (usual practice)

INTERVENTIONS:
Behavioral: Audit & feedback with educational outreach and facilitation — As in arm descriptions
  Arms: Audit & feedback with educational outreach and facilitation
Behavioral: Simple audit & feedback (usual practice) — As in arm descriptions
  Arms: Simple audit & feedback

SUMMARY:
In Canada, injury leads to more potential years of life lost and to greater costs than heart and stroke diseases combined. Furthermore, more than 50% of patients hospitalised following injury do not receive optimal care, 20% of injury deaths are estimated to be preventable, and significant variations in injury mortality and morbidity have been observed across trauma centers in Canada, the United Kingdom, Australia and the United States. Over the past decades, emphasis on adherence to evidence-based processes of care (rewards for doing more) and rapid innovation in imaging and therapeutic techniques has led to an exponential rise in unnecessary tests and procedures. Whole body computed tomography scan for single-system trauma is just one example. Low-value clinical practices, defined as "the common use of a particular intervention when the benefits don't justify the potential harm or cost" consume up to 30% of healthcare budgets. They expose patients to physical and psychological adverse events and put enormous pressure on healthcare budgets, thereby threatening accessible, universal health care. The objective of this research project is to evaluate the effectiveness of an intervention targeting reductions in low-value clinical practices for injury admissions. The results of this study should directly lead to improvements in the health systems across Canada and elsewhere. Medium and long-term advantages include an increase in healthcare efficiency and effectiveness, a reduction in costs, an increase in the availability of resources for patients who need them and a reduction in adverse events for patients hospitalized following injury.

DETAILED DESCRIPTION:
RATIONALE: While simple Audit & Feedback (A&F) has shown modest effectiveness for reducing low-value care, there is a knowledge gap on the effectiveness of multifaceted interventions to support de-implementation efforts. Given the need to make rapid decisions in a context of multiple diagnostic and therapeutic options, trauma is a high-risk setting for low-value care. Furthermore, trauma systems are a favorable setting for de-implementation interventions as they have quality improvement teams with medical leadership, routinely collected clinical data, and performance linked to accreditation.

OBJECTIVES: We aim to evaluate the effectiveness of a multifaceted intervention for reducing low-value clinical practices in acute adult trauma care.

METHODS: We will conduct a pragmatic cluster randomized controlled trial. Level I-III trauma centers in an inclusive Canadian trauma system (n=29) will be randomized (1:1) to receive simple A&F (control) or a multifaceted intervention (intervention). The multifaceted intervention, developed using extensive background work and United Kingdom Medical Research Council guidelines for the Development of Complex Interventions, includes an A&F report, educational materials, virtual educational meetings, and virtual facilitation visits. The primary outcome will be patient-level use of low-value initial diagnostic imaging, assessed using routinely collected trauma registry data. Secondary outcomes will be low-value specialist consultation, low-value repeat imaging for transfers, unintended consequences, and Incremental Cost-Effectiveness Ratios.

IMPACT: This innovative, timely research project will advance knowledge on the incremental effectiveness of a multifaceted intervention over simple A&F to de-implement low-value care. The intervention has a high probability of success because it targets a problem identified by stakeholders, is based on extensive background work, is low-cost, and is linked to accreditation. This intervention has the potential to reduce the adverse effects and indirect expenses of low-value trauma care for patients and families. It could also free up resources, reduce delays to care, and decrease healthcare professionals' workload, at a time of unprecedented strain on healthcare resources.

ELIGIBILITY:
Inclusion Criteria: All adult level I-III trauma centers in the Trauma Care Continuum of the province of Québec -

Exclusion Criteria: Level IV centers (patient volume too low)

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Low-value initial diagnostic imaging | 18-month interval (6 to 24 months) after implementation
  Proportion of low-risk patients who receive head, cervical spine or whole-body computed tomography in the emergency department

SECONDARY OUTCOMES:
Low-value specialist consultation | 18-month interval (6 to 24 months) after implementation
  Proportion of low-risk patients who receive neurosurgical or spine surgery consultation
Pre-transfer imaging | 18-month interval (6 to 24 months) after implementation
  Proportion of patients with a clear indication to transfer who receive imaging in referral center
Repeat post-transfer imaging | 18-month interval (6 to 24 months) after implementation
  Proportion of patients with imaging in referral center with no disease progression who are re-imaged in receiving center following transfer

OTHER OUTCOMES:
Mortality | 18-month interval (6 to 24 months) after implementation
  Proportion of patients admitted who die in hospital
Unplanned readmission | 18-month interval (6 to 24 months) after implementation
  Proportion of patients discharged alive with an unplanned readmission within 30 days of discharge
Missed injuries | 18-month interval (6 to 24 months) after implementation
  Proportion of patients admitted for whom an injury was missed in the emergency department and later detected as an inpatient
Hospital stay | 18-month interval (6 to 24 months) after implementation
  Mean hospital length of stay in days for all hospital admissions
Intensive care unit stay | 18-month interval (6 to 24 months) after implementation
  Mean intensive care unit stay in days for all patients admitted to the intensive care unit
Complications | 18-month interval (6 to 24 months) after implementation
  Proportion of patients admitted with an event of deep vein thrombosis/pulmonary embolism, decubitus ulcers, delirium, pneumonia, or urinary tract infection during their in-patient stay
Incremental Cost-Effectiveness Ratios | 0 to 24 months after implementation
  Economic evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data are held by provincial authorities and cannot be transmitted by study investigators. Supporting material will be made available through the study program website.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Six months after publication of all study results up to 10 years after study initiation
Access Criteria: Supporting data will be made available on request. Patient-level data from the provincial trauma registry can be accessed on request through provincial authorities.

REFERENCES:
- [Background] Moore L, Berube M, Tardif PA, Lauzier F, Turgeon A, Cameron P, Champion H, Yanchar N, Lecky F, Kortbeek J, Evans D, Mercier E, Archambault P, Lamontagne F, Gabbe B, Paquet J, Razek T, Stelfox HT; Low-Value Practices in Trauma Care Expert Consensus Group. Quality Indicators Targeting Low-Value Clinical Practices in Trauma Care. JAMA Surg. 2022 Jun 1;157(6):507-514. doi: 10.1001/jamasurg.2022.0812. PMID 35476055
- [Background] Moore L, Berube M, Tardif PA, Lauzier F, Turgeon A, Cameron P, Champion H, Yanchar N, Lecky F, Kortbeek J, Evans D, Mercier E, Archambault P, Lamontagne F, Gabbe B, Paquet J, Razek T, Belcaid A, Berthelot S, Malo C, Lang E, Stelfox HT. Validation of Quality Indicators Targeting Low-Value Trauma Care. JAMA Surg. 2022 Sep 14;157(11):1008-16. doi: 10.1001/jamasurg.2022.3912. Online ahead of print. PMID 36103195
- [Background] Moore L, Lauzier F, Tardif PA, Boukar KM, Farhat I, Archambault P, Mercier E, Lamontagne F, Chasse M, Stelfox HT, Berthelot S, Gabbe B, Lecky F, Yanchar N, Champion H, Kortbeek J, Cameron P, Bonaventure PL, Paquet J, Truchon C, Turgeon AF; Canadian Traumatic brain injury Research Consortium. Low-value clinical practices in injury care: A scoping review and expert consultation survey. J Trauma Acute Care Surg. 2019 Jun;86(6):983-993. doi: 10.1097/TA.0000000000002246. PMID 31124896
- [Background] Soltana K, Moore L, Bouderba S, Lauzier F, Clement J, Mercier E, Krouchev R, Tardif PA, Belcaid A, Stelfox T, Lamontagne F, Archambault P, Turgeon A; Canadian Traumatic Brain Injury Research Consortium. Adherence to Clinical Practice Guideline Recommendations on Low-Value Injury Care: A Multicenter Retrospective Cohort Study. Value Health. 2021 Dec;24(12):1728-1736. doi: 10.1016/j.jval.2021.06.008. Epub 2021 Aug 18. PMID 34838270
- [Background] Abiala G, Berube M, Mercier E, Yanchar N, Stelfox HT, Archambault P, Bourgeois G, Belcaid A, Neveu X, Isaac CJ, Clement J, Lamontagne F, Moore L. Pre- and posttransfer computed tomography imaging in Canadian trauma centers: A multicenter retrospective cohort study. Acad Emerg Med. 2022 Sep;29(9):1084-1095. doi: 10.1111/acem.14536. Epub 2022 Jun 8. PMID 35612384
- [Background] Moore L, Tardif PA, Lauzier F, Berube M, Archambault P, Lamontagne F, Chasse M, Stelfox HT, Gabbe B, Lecky F, Kortbeek J, Lessard Bonaventure P, Truchon C, Turgeon AF. Low-Value Clinical Practices in Adult Traumatic Brain Injury: An Umbrella Review. J Neurotrauma. 2020 Dec 15;37(24):2605-2615. doi: 10.1089/neu.2020.7044. Epub 2020 Sep 30. PMID 32791886
- [Background] Berube M, Moore L, Tardif PA, Berry G, Belzile E, Lesieur M, Paquet J. Low-value injury care in the adult orthopaedic trauma population: A systematic review. Int J Clin Pract. 2021 Dec;75(12):e15009. doi: 10.1111/ijcp.15009. Epub 2021 Nov 30. PMID 34816530
- [Derived] Berube M, Lapierre A, Sykes M, Grimshaw J, Turgeon AF, Lauzier F, Taljaard M, Stelfox HT, Witteman H, Berthelot S, Mercier E, Gonthier C, Paquet J, Fowler R, Yanchar N, Haas B, Lessard-Bonaventure P, Archambault P, Gabbe B, Guertin JR, Ouyang Y, Moore L; Canadian Traumatic Brain Injury Research Consortium. Development and usability testing of a multifaceted intervention to reduce low-value injury care. BMC Health Serv Res. 2025 Jan 7;25(1):37. doi: 10.1186/s12913-024-12153-y. PMID 39773251
- [Derived] Moore L, Berube M, Belcaid A, Turgeon AF, Taljaard M, Fowler R, Yanchar N, Mercier E, Paquet J, Stelfox HT, Archambault P, Berthelot S, Guertin JR, Haas B, Ivers N, Grimshaw J, Lapierre A, Ouyang Y, Sykes M, Witteman H, Lessard-Bonaventure P, Gabbe B, Lauzier F; Canadian Traumatic Brain Injury Research Consortium (CTRC). Evaluating the effectiveness of a multifaceted intervention to reduce low-value care in adults hospitalized following trauma: a protocol for a pragmatic cluster randomized controlled trial. Implement Sci. 2023 Jul 7;18(1):27. doi: 10.1186/s13012-023-01279-y. PMID 37420284